CLINICAL TRIAL: NCT01112670
Title: The Role of P-glycoprotein in Sitagliptin Clinical Pharmacology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 09-0531; R03DK084089 (NIH)
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Sitagliptin Phosphate; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABCB1 Group 1 (Experimental): ABCB1 CGC/CGC genetic make-up; sitagliptin 100 mg x 1 dose; atorvastatin 40 mg x 5 doses
  Interventions: Drug: Sitagliptin; Drug: atorvastatin
- ABCB1 Group 2 (Experimental): ABCB1 CGC/TTT genetic make-up; sitagliptin 100 mg x 1 dose; atorvastatin 40 mg x 5 doses
  Interventions: Drug: Sitagliptin; Drug: atorvastatin
- ABCB1 Group 3 (Experimental): ABCB1 TTT/TTT genetic make-up; sitagliptin 100 mg x 1 dose; atorvastatin 40 mg x 5 doses
  Interventions: Drug: Sitagliptin; Drug: atorvastatin

INTERVENTIONS:
Drug: Sitagliptin — sitagliptin 100 mg x 1 dose
  Other Names: Januvia
Drug: atorvastatin — atorvastatin 40 mg x 5 doses
  Other Names: Lipitor

SUMMARY:
The purpose of this study is to determine the pharmacogenetics, pharmacokinetics, and drug-drug interactions of sitagliptin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 21 to 60 years of age will be recruited to participate in this study.
* Subjects will be eligible if metabolic, renal, hepatic, and hematological laboratory tests are within normal limits.

Exclusion Criteria:

* Subjects will be excluded from the study if they have a current or past history of cardiovascular, hepatic, endocrine (e.g., diabetes), renal, pancreatic, gastrointestinal, pulmonary, immunologic, hematologic, or neurologic disease.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Aquilante, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited from the Denver metro area between November 2009 and December 2010.
Pre-assignment Details: Participants (n=145) were genetically pre-screened for ABCB1 1236/2677/3435 diplotypes. Those who possessed the needed ABCB1 genetic diplotypes, along with requisite clinical inclusion criteria, were started in the study (n=33).
Groups:
- ABCB1 Group 1: ABCB1 CGC/CGC genetic make-up. Sitagliptin to Sitagliptin+Atorvastatin. 8 participants started. 7 participants completed.
- ABCB1 Group 1*: ABCB1 CGC/CGC genetic make-up. Sitagliptin+Atorvastatin to Sitagliptin. 3 participants started. 3 participants completed.
- ABCB1 Group 2: ABCB1 CGC/TTT genetic make-up. Sitagliptin to Sitagliptin+Atorvastatin. 7 participants started. 6 participants completed.
- ABCB1 Group 2*: ABCB1 CGC/TTT genetic make-up. Sitagliptin+Atorvastatin to Sitagiptin. 4 participants started. 4 participants completed.
- ABCB1 Group 3: ABCB1 TTT/TTT genetic make-up. Sitagliptin to Sitagliptin+Atorvastatin. 6 participants started. 5 participants completed.
- ABCB1 Group 3*: ABCB1 TTT/TTT genetic make-up. Sitagliptin+Atorvastatin to Sitagliptin. 5 participants started. 5 participants completed.
Period: Sitagliptin to Sitagliptin+Atorvastatin
Arm/Group | ABCB1 Group 1 | ABCB1 Group 1* | ABCB1 Group 2 | ABCB1 Group 2* | ABCB1 Group 3 | ABCB1 Group 3*
Started | 8 | 0 | 7 | 0 | 6 | 0
Completed | 7 | 0 | 6 | 0 | 5 | 0
Not Completed | 1 | 0 | 1 | 0 | 1 | 0
Period: Sitagliptin+Atorvastatin to Sitagliptin
Arm/Group | ABCB1 Group 1 | ABCB1 Group 1* | ABCB1 Group 2 | ABCB1 Group 2* | ABCB1 Group 3 | ABCB1 Group 3*
Started | 0 | 3 | 0 | 4 | 0 | 5
Completed | 0 | 3 | 0 | 4 | 0 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All participants who participated in at least one period of the study (n=33)
Arm/Group | Overall Study Population
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Sitagliptin Monotherapy: Sitagliptin Area Under the Plasma Concentration-time Curve (AUC) From 0 to Infinity
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Groups:
- ABCB1 Group 1: ABCB1 CGC/CGC genetic make-up
- ABCB1 Group 2: ABCB1 CGC/TTT genetic make-up
- ABCB1 Group 3: ABCB1 TTT/TTT genetic make-up
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ng*hr/ml | 3638 (1439) | 3502 (1133) | 3129 (795)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.83, ANOVA

2. Primary Outcome: Sitagliptin Monotherapy: Sitagliptin Maximum Plasma Concentration (Cmax)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ng/ml | 454 (180) | 438 (152) | 394 (160)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.67, ANOVA

3. Secondary Outcome: Sitagliptin + Atorvastatin: Sitagliptin Area Under the Plasma Concentration-time Curve (AUC) From 0 to Infinity
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ng*h/ml | 3501 (1617) | 3430 (1279) | 3117 (1216)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.90, ANOVA

4. Secondary Outcome: Sitagliptin + Atorvastatin: Sitagliptin Maximum Plasma Concentration (Cmax)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- ABCB1 Group 2: ABCB1 CGC/CGC genetic make-up
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ng/ml | 428 (201) | 420 (137) | 370 (217)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.56, ANOVA

5. Other Pre Specified Outcome: Relative Change in Sitagliptin Area Under the Plasma Concentration-time Curve (AUC) From 0 to Infinity
Description: AUC of sitagliptin when administered with atorvastatin divided by AUC of sitagliptin when administered alone
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ratio | 0.96 [0.81 to 1.11] | 0.98 [0.88 to 1.07] | 0.97 [0.87 to 1.08]
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.97, ANOVA

6. Other Pre Specified Outcome: Relative Change in Sitagliptin Maximum Plasma Concentration (Cmax)
Description: Cmax of sitagliptin when administered with atorvastatin divided by Cmax of sitagliptin when administered alone
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ratio | 0.96 [0.75 to 1.17] | 1.0 [0.79 to 1.21] | 0.93 [0.76 to 1.11]
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.86, ANOVA

7. Primary Outcome: Sitagliptin Monotherapy: Sitagliptin Renal Clearance (CLr)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study and who had complete urine data.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 7 | 9 | 10
ml/min | 254 (176) | 232 (62) | 359 (182)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.21, ANOVA

8. Secondary Outcome: Sitagliptin + Atorvastatin: Sitagliptin Renal Clearance (CLr)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 7 | 9 | 10
ml/min | 280 (124) | 226 (66) | 339 (188)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.22, ANOVA

9. Other Pre Specified Outcome: Relative Change in Sitagliptin Renal Clearance (CLr)
Description: CLr of sitagliptin when administered with atorvastatin divided by CLr of sitagliptin when administered alone
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 7 | 9 | 10
ratio | 1.22 [0.97 to 1.48] | 0.99 [0.82 to 1.16] | 1.0 [0.81 to 1.18]
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.14, ANOVA

10. Other Pre Specified Outcome: Atorvastatin Area Under the Plasma Concentration Time Curve (AUC) Over the Dosing Interval (0-24 Hours)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ng*h/ml | 44.4 (28.0) | 35.4 (35.6) | 49.0 (37.1)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.29, ANOVA

11. Other Pre Specified Outcome: Atorvastatin Maximum Plasma Concentration (Cmax)
Time Frame: 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed both periods of the pharmacokinetic crossover study.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | ABCB1 Group 1 | ABCB1 Group 2 | ABCB1 Group 3
Number analyzed (Participants) | 9 | 10 | 10
ng/ml | 8.6 (6.2) | 7.5 (7.6) | 10.6 (7.4)
Statistical Analysis 1: Comparison: ABCB1 Group 1 vs ABCB1 Group 2 vs ABCB1 Group 3; Test type: Superiority or Other; p = 0.43, ANOVA

ADVERSE EVENTS:
Time Frame: Pharmacokinetic study periods
Groups:
- Overall Study Population: All participants who started the study (n=33)
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 24/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Population (N=33)
Headache (General disorders) | 11 (11)
Lightheadedness (General disorders) | 3 (3)
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nasal congestion (General disorders) | 2 (2)
Increased liver function tests (Hepatobiliary disorders) | 3 (3)
Hypoalbuminemia (General disorders) | 8 (8)
Pain at IV site (General disorders) | 3 (3)
Dry mouth (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Findings are only applicable to individuals with ABCB1 CGC/CGC, CGC/TTT, or TTT/TTT diplotypes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No